CLINICAL TRIAL: NCT05197855
Title: Evolution of Sleep Quality During the Initiation of Continuous Positive Airway Pressure Treatment in Obstructive Sleep Apnea Syndrome: an Exploratory Study
Brief Title: Sleep Quality Evolution: Dreem Under CPAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Dreem (Industry); AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.0346
Record Dates: First submitted 2021-12-01; First posted 2022-01-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure (CPAP); Technological innovations; Sleep Stages; Dreem Headband
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Technological innovations and CPAP (Experimental): Patients will be equipped with 4 devices: a Dreem 3 Headband, a pulse oximeter, a continuous glucose sensor, and a pedometer. In parallel they will be equipped by the CPAP at home by Icadom.
  Interventions: Device: Deem 3 Headband

INTERVENTIONS:
Device: Deem 3 Headband — The patient will wear the Dreem 3 headband and pulse oximeter at home before initiation of CPAP (for 7 nights) and during a month of treatment (for a minimum of 9 nights), after the initiation of CPAP. He will also wear a glucose sensor and a pedometer during the entire study period before and after CPAP treatment.

SUMMARY:
Continuous positive airway pressure (CPAP) has a caricatural effect in reducing nocturnal respiratory abnormalities and improving the micro-and macrostructure of sleep. Studies characterizing the improvement of acute sleep parameters after the initiation of CPAP are limited to one or two nights of polysomnographic recording. This is related to the cost of performing these studies with repeated recordings in the laboratory and to the acceptability by patients to perform multiple nights of recordings.

Investigators currently have powerful and reliable methods allowing us to carry out nights at home in the patient's ecosystem, in real-life conditions. The characterization of sleep parameters by these methods is equivalent to a polysomnographic recording.

These technological innovations will allow us to characterize sleep before the initiation of CPAP treatment during several nights performed at home. Investigators will then be able to characterize the kinetics and stability of the improvement of sleep parameters in patients with obstructive sleep apnea syndrome in whom continuous positive airway pressure is initiated.

These data will be original and will serve as exploratory data to judge whether the objective improvement of sleep parameters in the first weeks of treatment is associated with improvement in sleepiness, quality of life, and compliance with treatment.

DETAILED DESCRIPTION:
This study aims to evaluate the quality of sleep, principally the deep slow-wave sleep (sleep stage N3) before and after the initiation of continuous positive airway pressure (CPAP) treatment.

70 newly diagnosed patients with OSA requiring CPAP treatment, will be included.

For the study, they will wear the Dreem 3 headband and pulse oximeter at home before initiation of CPAP (for 7 nights) and during the first month of CPAP (for a minimum of 9 nights). They will be also equipped with a glucose sensor and a pedometer during the entire study period before and after CPAP treatment.

Patients will also complete questionnaires about their health status before CPAP treatment (at inclusion) and after one month of treatment

These devices will allow the measurements of different parameters: sleep stages, total sleep time, sleep measures derived from sleep stages, snoring, breathing rate, heart rate head movements, arterial hemoglobin oxygen saturation, pulse rate, continuous subcutaneous glucose level, and physical activity data (average daily steps, average distance walked per day).

This will generate interesting data on the sleep parameters and their evolution during the initiation of the CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with OSA requiring CPAP treatment
* Patients able to use a mobile application on a smartphone or tablet
* Patients with access to a wi-fi internet connection at home
* Patients agreeing to remote monitoring of CPAP compliance data by the home care provider
* Patients who have signed consent to participate in the study
* Subjects affiliated to a social security

Exclusion Criteria:

* Patients already treated for OSA
* Patients treated with a sleep aid (sleeping medications)
* Patients with severe chronic obstructive or restrictive lung disease with or without oxygen
* Patients with unstable cardiovascular disease or severe heart failure requiring hospitalization within the last three months or meeting New York Heart Association criteria, Class III or IV disease
* Subjects listed in articles L1121-5 to L1121-8: pregnant women, feeding and parturients, subjects deprived of liberty by judicial or administrative decision, persons under legal protection
* Persons in a period of exclusion from another study or ongoing participation in a drug study
* Subjects likely, at the investigator's discretion, to be uncooperative or noncompliant with the obligations inherent to participation in the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Duration of deep slow-wave sleep (sleep stage N3) before and after initiation of continuous positive airway pressure (CPAP) treatment. | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Time spent on the deep slow-wave sleep stage (stage N3 sleep), recorded by the Dreem 3 headband, from 7 nights before and 9 nights after initiation of CPAP treatment

SECONDARY OUTCOMES:
Duration of the other sleep stages (W, N1, N2 and REM) | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Sleep stages (W, N1, N2 and REM) and total sleep time spent in each sleep stage, recorded by the Dreem 3. All the data units are in minutes
Duration of different sleep times | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Sleep parameters recorded by Dreem 3 headband: sleep times (bedtime, total sleep time (TST), sleep onset delay (SOD),time in bed (TIB), time awake after falling asleep (WASO), final wakefulness time)
The percentage of time while sleeping | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Sleep parameter recorded by Dreem 3 headband: sleep efficiency ((TST/TIB) x100)
The frequences of sleep waves during the NREM sleep stage recorded by Dreem 3 headband | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  sleep spindle density expressed in Hertz recorded by the EEG sensors
The frequence of snoring while sleeping recorded by Dreem 3 headband | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  snoring is expressed in decibel minute recorded by a microphone integrated in the Dreem3
Respiratory rate measurment recorded by Dreem 3 headband | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  It is expressed in breathe per minute recorded accelerometer sensor
Heart rate measurement while sleepingrecorded by Dreem 3 headband | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Expressed in beats per minute recorded by accelerometer sensor
The position of the head changes while sleeping recorded by Dreem 3 headband | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Head movements are recorded by an accelerometer sensor in the Dreem 3 Headband
Evolution of the nocturnal oximetry | 7 nights before CPAP initiation and for a month (minimum 9 nights) after CPAP initiation
  Nocturnal oxygen saturation measured by a pulse oximeter
Evolution of the subcutaneous glucose level | 7 nights before CPAP initiation and for a month after CPAP initiation
  Continuous subcutaneous glucose level (measured by FreeStyle Libre 2 continuous glucose sensor)
Evolution of glycemia | At inclusion and a month after CPAP initiation
  Blood glucose level by blood sampling
Average daily number of steps | 7 nights before CPAP initiation and for a month after CPAP initiation
  It will be measured by a Garmin Vivofit 3 pedometer expressed in steps/day
Average distance walked per day | 7 nights before CPAP initiation and for a month after CPAP initiation
  It will be measured by a Garmin Vivofit 3 pedometer expressed in Kilometer
Sleep quality assessed by Pittsburg questionnaire | At inclusion and a month after CPAP initiation
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Severity of insomnia measured by the index sverety of insomnia questionnaire | At inclusion and a month after CPAP initiation
  The general ISI score varies between 0 and 28: -7 = No insomnia 8-14 = Sub-clinical insomnia (mild) 15-21 = Clinical insomnia (moderate) 22-28 = Clinical insomnia (severe)
Evolution of the somnolence | At inclusion and a month after CPAP initiation
  Epworth Sleepiness Score (ESS):
  0 = no chance of dozing or falling asleep
  1. = low chance of falling asleep
  2. = medium chance of falling asleep
  3. = high chance of falling asleep
Evolution of the quality of life by the Short Form 36 health survey questionnaire | At inclusion and a month after CPAP initiation
  A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Evolution of the compliance of CPAP treatment | For a month during CPAP treatment
  Collection of average CPAP treatment use (in hours/day) provided by telemonitoring
Evolution of the effectiveness of CPAP treatment | For a month during CPAP treatment
  Collection of residual AHI provided by telemonitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pépin, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital (CHUGA)
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No